CLINICAL TRIAL: NCT03353831
Title: Atezolizumab in Combination With Bevacizumab and Chemotherapy Versus Bevacizumab and Chemotherapy in Recurrent Ovarian Cancer - a Randomized Phase III Trial
Brief Title: Atezolizumab With Bevacizumab and Chemotherapy vs Bevacizumab and Chemotherapy in Early Relapse Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Research GmbH (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGO-OVAR 2.29
Record Dates: First submitted 2017-11-14; First posted 2017-11-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Ovarian Carcinoma
Keywords: Recurrent Ovarian Cancer; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; atezolizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Chemotherapy + Bevacizumab + Placebo (Placebo Comparator): Chemotherapy: Paclitaxel 80 mg/m² d1, 8, 14, 22 q28 or pegylated liposomal doxorubicin 40 mg/m² q28 + Bevacizumab 10 mg/kg q14 + Placebos q14
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy; Drug: Placebos
- Arm B: Chemotherapy + Bevacizumab + Atezolizumab (Experimental): Chemotherapy: Paclitaxel 80 mg/m² d1, 8, 14, 22 q28 or pegylated liposomal doxorubicin 40 mg/m² q28 + Bevacizumab 10 mg/kg q14 + Atezolizumab 840 mg q14
  Interventions: Drug: Bevacizumab; Drug: Atezolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be administered by intravenouse route at a dose of 10mg/kg q14 during the treatment period
Drug: Atezolizumab — Atezolizumab will be administered by intravenous route at a dose of 840 mg q14 during the treatment period
  Arms: Arm B: Chemotherapy + Bevacizumab + Atezolizumab
Drug: Chemotherapy — Chemotherapy (Paclitaxel or PLD) will be administered by intravenous route at different doses during the treatment period q28
Drug: Placebos — Placebo will be administered by intravenous route q14 during the treatment period
  Arms: Arm A: Chemotherapy + Bevacizumab + Placebo

SUMMARY:
This is a phase III, randomized, partially blinded, multicenter trial to evaluate the efficacy and safety of atezolizumab plus bevacizumab and chemotherapy compared to placebo plus bevacizumab and chemotherapy in patients with recurrent ovarian-, fallopian tube, or primary peritoneal cancer with 1st or 2nd relapse within 6 months after platinum based chemotherapy or 3rd relapse.

DETAILED DESCRIPTION:
Approximately 550 patients will be randomized in a 1:1 ratio to the treatments as specified below:

Arm A: Chemotherapy + Bevacizumab + Placebo Arm B: Chemotherapy + Bevacizumab + Atezolizumab

Study treatment will continue until disease progression per RECIST v1.1, unacceptable toxicity, or patient or investigator decision to discontinue treatment. Atezolizumab/placebo, chemotherapy and bevacizumab may be discontinued for toxicity independently of each other in the absence of disease progression.

For each patient, chemotherapy (PLD or Paclitaxel weekly) will be selected by the investigator prior to randomization.

Recruitment to an individual chemotherapy cohort will be closed once 50% of patients are recruited to this cohort. In such case the remaining cohort will remain open for recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically diagnosed ovarian, fallopian tube, or primary peritoneal cancer
2. Relapsed disease
3. Patients with up to three prior therapies. In patients with 1 or 2 prior treatment lines, the treatment free interval after platinum has to be less than 6 months; in addition patients with three prior lines of chemotherapy who are not considered for platinum-containing chemotherapy lines are also eligible
4. Measurable disease, evaluable disease in combination with GCIG CA-125 criteria, or histologically proven relapse/progression
5. Mandatory de novo tumor biopsy (not older than 3 months) sent to central laboratory as formalin-fixed, paraffin-embedded (FFPE) sample for determination of PDL1 status prior to randomization for stratification.
6. Availability of a representative archival FFPE tumor sample (preferable from primary diagnosis)
7. Patient has not progressed on the chosen/planned chemotherapy (PLD or Paclitaxel) in any prior line
8. Patients previously treated with bevacizumab are eligible, with the exclusion of those patients that has suspended bevacizumab for more than 2 subsequent cycles or permanently discontinued bevacizumab during their previous treatment due to toxicity.
9. Females aged ≥ 18 years at signing at time of signing informed consent form
10. Signed written informed consent and ability to comply with the study protocol, in the investigator's judgement
11. Adequate hematological, renal and hepatic function within 28 days prior to first administration of study treatment:

    * Hemoglobin ≥ 9.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.5 x 10xE^9/L
    * Platelet count ≥ 100 x 10xE^9/L
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT) ≤ 2.5 x ULN, unless liver metastases are present, in case of liver metastases values must be ≤ 5 x ULN
    * Serum creatinine ≤ 1.5 x institutional ULN
    * Patient not receiving anticoagulant medication who has an International Normalized Ratio (INR) ≤ 1.5 and an Activated ProThrombin Time (aPTT) ≤ 1.5 x ULN. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to site medical standard). If the patient is on oral anticoagulants, dose has to be stable for at least two weeks at the time of randomization
    * Urine dipstick for proteinuria < 2+. If urine dipstick is ≥ 2+, 24-hours urine must demonstrate ≤ 1 g of protein in 24 hours.
12. Patients must have adequately controlled blood pressure (BP), with a systolic BP of ≤ 140 mmHg and diastolic BP of ≤ 90 mmHg for eligibility. Patients must have a BP of ≤ 140/90 mmHg taken in the clinic setting by a medical professional within 2 weeks prior to starting study.
13. Estimated life expectancy of at least 3 months
14. ECOG performance status 0 - 1
15. Negative urine or serum pregnancy test within 7 days of study treatment in women of childbearing potential (WOCBP), confirmed prior to treatment on day 1
16. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 5 months after administration of the last dose of atezolizumab/placebo and 6 months after the last dose of bevacizumab, paclitaxel, or PLD, whichever is later.
17. For countries where this will apply to: a patient will be eligible for randomization in this study only, if either affiliated to, or a beneficiary of a social security category.
18. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, that include the completion of patient-reported outcomes questionnaires.

Exclusion Criteria:

1. Non-epithelial tumor origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors)
2. Ovarian tumors of low malignant potential (e.g. borderline tumors)
3. Malignancies other than ovarian cancer within 5 years prior to randomisation, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%) and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, non melanoma skin carcinoma, ductal carcinoma in situ, or Stage I uterine cancer)
4. More than three prior systemic anticancer regimens; maintenance therapies (e.g. with bevacizumab, olaparib or niraparib) are not calculated as separate line.
5. Prior systemic anticancer therapy within 28 days before randomization (except bevacizumab: 20 days).
6. Prior radiotherapy to the pelvis or the abdomen.
7. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement thera-py is permitted).
8. Prior treatment with anti-CD137 or immune checkpoint blockade therapies, anti-PD1, or anti-PD-L1 therapeutic antibodies or anti-CTLA 4
9. Prior randomization in AGO-OVAR 2.29.
10. Treatment with systemic immunostimulatory agents (in-cluding but not limited to interferon-alpha (IFN-α) and interleukin-2 (IL-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to cycle 1, day 1.
11. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophos-phamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor [TNF] agents) within 2 weeks prior to cycle 1, day 1, or anticipated requirement for systemic immunosuppressive medications during the trial.

    The use of inhaled corticosteroids for chronic obstruc-tive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
12. Patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have screening and subsequent tumor assessments performed using magnetic resonance imaging (MRI).
13. Administration of a live, attenuated vaccine within 4 weeks prior to cycle 1, day 1 or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after the last dose of atezolizumab/placebo. Influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccination
14. Major surgery within 4 weeks of starting study treatment or patient who has not completely recovered from the effects of any major surgery. Core biopsy or other minor surgical procedure within 7 days prior to day 1, cycle 1 is permitted.
15. Previous allogeneic bone marrow transplant or previous solid organ transplantation.
16. Current treatment with anti-viral therapy for HBV.
17. History of idiopathic pulmonary fibrosis (including pneumonitis), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evi-dence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) detected on screening chest CT scan is permitted
18. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to randomization
19. History or evidence hemorrhagic disorders within 6 months prior to randomization
20. Patients are excluded if having a history or evidence of thrombosis as follows:

    * Any Grade 4 thrombosis
    * Arterial thrombosis within 6 months prior to ran-domization
    * Grade ≤ 3 venous thrombosis within 3 months prior to randomization Patients with central venous access thrombosis are eligi-ble.
21. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of sus-pected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of sus-pected spinal cord compression
22. History of autoimmune disease, including but not limited to dermatomyositis, myasthenia gravis, myositis, auto-immune hepatitis, systemic lupus erythematosus, rheu-matoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guil-lain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Except patients with:

    * a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone
    * controlled type 1 diabetes mellitus on a stable insulin regimen

    Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
23. Any prior history of hypertensive crisis (CTCAE grade 4) or hypertensive encephalopathy.
24. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    Patients with past hepatitis B virus (HBV) infection or re-solved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
25. Persistent toxicities (≥ CTCAE grade 2) with the exception of alopecia, caused by previous cancer treatment. Neurotoxicity CTCAE grade 2 is permitted in case the patient is planned for PLD treatment.
26. Severe infection requiring oral or IV antibiotics within 4 weeks prior to randomization, including but not limited to active tuberculosis or hospitalization for complications of infection, bacteremia, or severe pneumonia. Patients receiving prophylactic antibiotics (e.g., to prevent urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
27. Current or recent (within 10 days prior randomization) chronic use of aspirin > 325 mg/day.
28. Clinically significant (e.g. active) cardiovascular disease, including:

    * Myocardial infarction or unstable angina pectoris within ≤ 6 months of randomization
    * New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF)
    * Poorly controlled cardiac arrhythmia despite medica-tion (patients with rate controlled atrial fibrillation are eligible)
    * Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision)
    * Resting ECG with QTc >470 msec or family history of long QT syndrome
29. For patients with PLD treatment: Left ventricular ejection fraction defined by ECHO below the institutional lower limit of normal
30. Evidence of bleeding diathesis or significant coagulopathy (in the absence of anticoagulation).
31. Non-healing wound, active ulcer or bone fracture.
32. History of bowel obstruction (including subocclusive disease) related to underlying disease, a history of ab-dominal fistula, GI perforation, or intra-abdominal abscess, or evidence of deep infiltration of the bowel by pelvic examination or on computed tomography, or clinical symptoms of bowel obstruction.
33. Patients with evidence of abdominal free air.
34. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications
35. Known hypersensitivity or allergy to drugs containing Chinese hamster (CHO) ovary cells or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
36. Known hypersensitivity reaction or allergy to drugs chemically related to bevacizumab, paclitaxel, pegylated liposomal doxorubicin, or their excipients that contra-indicates the subject's participation.
37. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. This includes also any psychiatric disorder that prohibits obtaining informed consent.
38. Pregnancy, lactation, or intention to become pregnant during the study or within 5 months after the last dose of atezolizumab/placebo as well as breastfeeding women or intended to breastfeed during the study and up to 6 months after treatment with paclitaxel, bevacizumab and pegylated liposomal doxorubicin (PLD).
39. For France only: Patients deprived of their liberty by judicial or administrative decision and patients under a legal protection measure or unable to express their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of randomizationrandomization to date of death from any cause assessed up to 40 months
  regular patient contacts during the trial regarding life status
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs earlier, assessed up to 40 months
  Progressive Disease based on investigator assessment using RECIST v1.1

SECONDARY OUTCOMES:
patient reported outcomes (QLQ and PRO-CTCAE) | every 4 weeks during the first 3 months, then every 12 weeks until PD#1, assessed up to 40 months
  questionnaires to be completed by patients and collected frequently during the trial
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs earlier, assessed up to 40 months
  based on investigator assessment using RECIST v1.1
Duration of Response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs earlier, assessed up to 40 months
  based on investigator assessment using RECIST v1.1
Efficacy regarding PD-L1 status | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs earlier, assessed up to 40 months
  Efficacy regarding PD-L1 positivity defined by the VENTANA SP142 assay (negative: IC 0 versus positive IC: 1/2/3)

OTHER OUTCOMES:
Time from randomization to first subsequent therapy (TFST) | at every visit during the trial up to a maximum of 40 months
  time to first subsequent therapy
Time from randomization to second subsequent therapy (TSST) | at every visit during the trial up to a maximum of 40 months
  Time to second subsequent therapy
Analysis on LDH levels at baseline | Baseline
  normal vs. elevated values

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, MD, PhD, Study Chair — Kliniken Essen-Mitte, Germany
Locations (111):
- Medizinische Universität, Innsbruck, Austria
- Belgium (5):
  - UZA Edegem, Edegem
  - AZ Sint Lucas, Ghent
  - UZ Leuven, Leuven
  - CHU Liège Sart Tilman Grivegnée, Liège
  - CHU UCL Namur Sainte Elisabeth, Namur
- Denmark (4):
  - Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- East Tallinn Central Hospital, Tallinn, Estonia
- Tampere University Hospital, Tampere, Finland
- France (27):
  - ICO d'Angers, Angers
  - Institut Sainte Catherine, Avignon
  - Hôpital Jean Minjoz, Besançon
  - Blois Hospital (Centre Hospitalier de Blois), Blois
  - Clinique TIVOLI-DUCOS, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Médipôle de Savoie, Challes-les-Eaux
  - SASU Centre d'Oncologie et Radiothérapie 37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille, Lille
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - ORACLE Centre d'Oncologie de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Institut Curie Site Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Foch, Suresnes
  - IUCT Oncopole - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Germany (42):
  - Hochtaunus-Kliniken, Bad Homburg
  - Charité - Universitätsmedizin Berlin (CVK), Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Universitätsfrauenklinik Köln, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen-Mitte, Essen
  - Universitätsfrauenklinik Essen, Essen
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsfrauenklinik Frankfurt, Frankfurt
  - Klinikum Gütersloh, Gütersloh
  - Universitätsfrauenklinik Halle/Saale, Halle
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Praxisgemeinschaft Frauenärzte am Bahnhofsplatz, Hildesheim
  - Universitätsklinikum Jena, Jena
  - ViDia Christliche Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Universitätsfrauenklinik Mannheim, Mannheim
  - Johannes Wesling Klinikum, Minden
  - Klinikum der Universität München, München
  - Rotkreuzklinikum München, München
  - Universitätsklinikum Münster, Münster
  - MVZ Nordhausen, Nordhausen
  - Ortenau Klinikum Offenburg-Gengenbach, Offenburg
  - Onkologie Ravensburg, Ravensburg
  - Universitätsfrauenklinik Regensburg, Regensburg
  - Thüringen Kliniken "Georgius Agricola", Saalfeld
  - CTS CaritasKlinikum Saarbrücken, Saarbrücken
  - Leopoldina-Krankenhaus, Schweinfurt
  - Klinikum Traunstein, Traunstein
  - Universitätsfrauenklinik Tübingen, Tübingen
  - Universitätsfrauenklinik Ulm, Ulm
  - Helios Dr. Horst Schmidt Kliniken, Wiesbaden
  - Marien-Hospital, Witten
  - AMO MVZ Wolfsburg, Wolfsburg
- Lithuania (2):
  - Vilniaus universiteto ligoninė Santaros klinikos, Kaunas
  - Nacionalinis vėžio institutas, Vilnius
- Oslo University Hospital, Oslo, Norway
- Spain (16):
  - Hospital Clínic de Barcelona, Barcelona
  - Institut Català d'Oncologia (ICO) d'Hospitalet, Barcelona
  - Vall d'Hebron Instituto de Oncología (VHIO), Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Institut Català d'Oncologia (ICO) de Girona, Girona
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Hospital Universitario La Paz, La Paz
  - Clínica Universidad de Navarra (CUN), Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Son Llàtzer, Palma de Mallorca
  - Clínica Universidad de Navarra (CUN), Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Clínico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología (IVO), Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Malmo
  - Karolinska University Hospital, Solna
- Switzerland (8):
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Frauenfeld, Frauenfeld
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harter P, Marme F, Redondo A, Reuss A, Lindemann K, Kurzeder C, Van Nieuwenhuysen E, Marth C, Pietzner K, Ray-Coquard I, Garcia-Duran C, Jonuskiene G, Heitz F, Bellier C, Perez-Fidalgo JA, El-Balat A, Selle F, Romero I, Wimberger P, Follana P, Pardo B, de Gregorio N, Joly F, Gaba L, Burges A, Fabbro M, Hasenburg A, Fehm T, Schmalfeldt B, Pautier P. Atezolizumab With Bevacizumab and Nonplatinum Chemotherapy for Recurrent Ovarian Cancer: Final Results From the Placebo-Controlled AGO-OVAR 2.29/ENGOT-ov34 Phase III Trial. J Clin Oncol. 2026 Jan 10;44(2):103-116. doi: 10.1200/JCO-25-01210. Epub 2025 Dec 3. PMID 41337696
- [Derived] Harter P, Pautier P, Van Nieuwenhuysen E, Reuss A, Redondo A, Lindemann K, Kurzeder C, Petru E, Heitz F, Sehouli J, Degregorio N, Wimberger P, Burges A, Cron N, Ledermann J, Lorusso D, Paoletti X, Marme F. Atezolizumab in combination with bevacizumab and chemotherapy versus bevacizumab and chemotherapy in recurrent ovarian cancer - a randomized phase III trial (AGO-OVAR 2.29/ENGOT-ov34). Int J Gynecol Cancer. 2020 Dec;30(12):1997-2001. doi: 10.1136/ijgc-2020-001572. Epub 2020 Jun 30. PMID 32606097